CLINICAL TRIAL: NCT03390335
Title: Development of Decompression Tables for Diving at Altitude
Brief Title: Decompression Tables for Diving at Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro00087803
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Decompression Sickness; Acute Mountain Sickness
MeSH Terms: conditions — Decompression Sickness; Altitude Sickness | interventions — Pressure

STUDY DESIGN:
Intervention Model Description: This design is a two factor, incomplete block design - three altitudes (8,000, 10,000, and 12,000 feet) and 2 breathing gases (air, 35% O2-N2). The investigators expect to see 0 events in the combinations tested, calculated by the Bayesian Method. If the rate of events is larger than expected, the investigators will use logistic regression to assess if the main effect Air (Air vs. 35% O2-N2) or altitude (8,000, 10,000 or 12,000 feet) or the interaction of these 2 factors imparts relative increased risk. The investigators will set a Type-I error rate of 0.05 (two-tailed).In the presence of 'zero cells', the investigators will either (1) collapse cells into reasonable groups, or (2) add a very small set of constants to the frequency and assess the impact on the effect sizes and tests of significance.1 In the absence of an interaction effect, main effects will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Altitude Dive Altitude profile (Experimental): Subjects are exposed to Pressure profiles (Altitude followed by a Dive with a return to Altitude) and Breathing Gases during dive exposures.
  Interventions: Other: Pressure; Other: Breathing Gas

INTERVENTIONS:
Other: Pressure — Subjects undergo altitude exposure, diving exposure, and return to altitude. Altitudes: 8,000, 10,000, 12,000, or 15,000 feet Dives: 60 or 100 feet of sea water
Other: Breathing Gas — Subjects will breathe air, 35% Oxygen, Balance Nitrogen, or 100% Oxygen during the diving exposure

SUMMARY:
The aims of this proposal are to test current USN procedures for adjusting decompression procedures during air diving at 8,000 and 10,000 ft altitude and to provide a decompression algorithm for no-stop dives to 100 feet of sea water (fsw) at 10,000 and 12,000 ft altitude using enriched O2 (PO2=1.3 ATM). Additionally, the experiments will determine whether a period of hyperbaric hyperoxia, such as would be experienced during a dive at altitude, reverses altitude acclimatization, resulting in a return of acute mountain sickness (AMS) symptoms.

DETAILED DESCRIPTION:
Three different types of experiments will be performed:

(A). Testing of Cross corrections breathing air at 8,000 (0.743 ATA) and 10,000 ft (0.688 ATA). Subjects will be decompressed in a hypobaric chamber to one of the altitudes above. A no-stop dive to 60 fsw will be tested at each altitude (2.82 ATA at sea level, 2.56 ATA at 8,000 ft, 2.51 ATA at 10,000 ft). Using the Cross corrections, the virtual depth for both altitudes is 90 fsw, for which the no-stop time is 30 minutes. During the dive the subject will be immersed/submersed at rest/mild exercise in 28°C water. Ascent rate will be 30 fsw/min. Upon surfacing the diver will be monitored for 12 hours for symptoms of decompression sickness and transthoracic echocardiography (rest and leg/arm motion) to examine for venous gas embolism (VGE) at 5, 15, 30, 60 and 120 minutes after surfacing. After that, measurements will be continued until no bubbles are detected.

(B). Testing of a no-stop dive to 100 fsw at 10,000 ft and 12,000 ft breathing 35% O2. For this series of experiments all subjects will remain at altitude for 48 hours before diving, in order to allow for resolution of AMS symptoms. Appropriate depth-time profiles have been assessed by calculating the equivalent sea level air depth for each of these dives (PN2 values 2.42 and 2.36 ATM, respectively). These yield equivalent air depths of 68 and 66 fsw, respectively. Cross corrected virtual depths would therefore be 99 and 104 fsw, yielding no-stop times of 25 and 20 minutes, respectively. The Cross correction method will be used in this instance because, although largely untested, it is presently in use by the Navy. As with the air dives described above, the more provocative dives (12,000 ft) will be completed before the ones at 10,000 ft, which will increase the confidence for the bottom time used at the lower altitude.

(C). Testing to determine whether a high PO2 dive would reverse altitude acclimatization and re-establish susceptibility to AMS. Subjects will ascend in the chamber to 15,000 ft in a graded fashion over 12 hours (15,000 ft has been chosen due to extensive Duke experience with this altitude). Then, after 48 hours they will simulate a hyperoxic dive by breathing 100% O2 for 120 minutes at 1.3 ATA. This will simulate, for example, a 2 hour dive at 12,000 ft to 65 fsw breathing 50% O2. The diver will then return to 15,000 ft and remain at that altitude for 24 hours to allow for AMS symptoms to recur (if indeed they do). Lake Louise AMS scores will be collected every 8 hours. AMS symptoms will be treated with acetaminophen, NSAIDs and anti-emetics as needed. Subjects will be assessed clinically every 12 hours for high altitude pulmonary edema (HAPE) and high altitude cerebral edema (HACE). Occurrence of either HAPE or HACE will require that the subject be returned immediately to 1 ATA and treated appropriately.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* smoking, cardiorespiratory disease (including hypertension, airways obstruction), seizure disorder, pregnancy, history of middle ear or sinus disease or high altitude cerebral or pulmonary edema (HACE, HAPE), inability to perform middle ear autoinflation, anemia, sickle cell disease and sickle cell trait. Individuals with VO2peak <35 mL.kg-1.min-1 (males) and <30 mL.kg-1.min-1 (females)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Decompression Sickness | 12 hours
  Subjects will be evaluated for symptoms of decompression sickness when returning to the initial altitude following a dive exposure.
Maximum Acute Mountain Sickness (AMS) Score Change | 48 hour, 72 hours
  Lake Louise Scoring System for Acute Mountain Sickness. Subjects will fill out a six-question questionnaire (0 - 3, higher scores are worse symptoms) and a three-question clinical assessment (0-4, 0-4, 0-2, higher score is worse a assessment). The total score of all questions and assessments (0 - 28, higher is worse AMS), is determined every eight hours for 48 hours at altitude pre-dive and 24 hours at altitude post-dive.

SECONDARY OUTCOMES:
Venous Gas Emboli | 12 hours
  2D ultrasound will be used to assess right ventricular bubble score at 5, 15, 30, 60 and 120 minutes and hourly until no bubbles are detected using the following scale: Modified Eftedal-Brubakk Scale for Venous Gas Embolism (VGE)
  Grade Definition 0 No observable bubbles
  1. Occasional bubbles
  2. At least 1 bubble every 4 heart cycles
  3. At least 1 bubble every heart cycle
  4. A Continuous bubbling, 1-2 bubbles per cm2 in every image
  4B Continuous bubbling, at least 3 bubbles per cm2 in every image 4C Almost complete whiteout in the right heart, individual bubbles can still be discerned 5 "White out", single bubbles cannot be discriminated

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moon, MD, Principal Investigator — Duke Universtiy Health System
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No